CLINICAL TRIAL: NCT01018927
Title: Role of Cardiac MR (CMR) In Detecting Features of Early Myocardial Infiltration With Amyloid and Light Chain Deposition Disease in Subjects With Multiple Myeloma
Brief Title: Detecting Early Myocardial Infiltration w/Amyloid & Light Chain Deposition Disease in Multiple Myeloma Subjects
Status: Terminated | Type: Observational
Why Stopped: PI does not have time to continue study
Sponsor: University of Arkansas (Other)
Collaborators: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: 110104
Record Dates: First submitted 2009-11-16; First posted 2009-11-25 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: Cardiac MR (CMR); Early Myocardial Infiltration; Amyloid; Light Chain Deposition Disease; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Additional MRI images: Prospective review of 100 CMR studies performed on multiple myeloma patients referred for cardiac evaluation by MRI. Three additional MRI images will be performed to determine the role of cardiac MR (CMR) in detecting features of early myocardial infiltration
  Interventions: Device: Administering three additional MRI images

INTERVENTIONS:
Device: Administering three additional MRI images — Three additional MRI images to determine the role of cardiac MR (CMR) in detecting features of early myocardial infiltration

SUMMARY:
The purpose of this study is to see if MRI techniques can be used for early evaluation of cardiac amyloidosis which is sometimes seen in individuals with multiple myeloma. Cardiac amyloidosis is a medical disorder that decreases heart function.

DETAILED DESCRIPTION:
The purpose is to investigate the use of multiple newer CMR techniques for early evaluation of cardiac amyloidosis in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* All races and ethnic groups
* Male and female ages 18-80 years of age
* History of multiple myeloma
* CMR study for evaluation for cardiac amyloidosis

Exclusion Criteria:

* Pregnant women
* Subject with a metallic or electronic or other device that could be affected by the magnet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma subjects
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2009-06; Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
This study is to see if MRI techniques can be used for early evaluation of cardiac amyloidosis which is sometimes seen in individuals with multiple myeloma. | The time frame is five additional minutes & three additional images during and MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Pandey, Principal Investigator — University of Arkansas for Medical Sciences (UAMS)
Locations (1):
- University or Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas, United States